CLINICAL TRIAL: NCT01151007
Title: Study of KRAS Mutation in 250 Cases of Colorectal Carcinoma and Study of the Incidence of the Disease in Martinique, From 2007 to 2009
Brief Title: KRAS Mutation and Incidence of the Colorectal Carcinoma in Martinique Between 2007 and 2009
Acronym: KRAS
Status: Completed | Type: Observational
Sponsor: University Hospital Center of Martinique (Other)
Responsible Party: Sponsor
Other Study IDs: 10/E/11
Record Dates: First submitted 2010-06-24; First posted 2010-06-25 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Colorectal Carcinoma
Keywords: Kras mutation; colorectal carcinoma; Martinique
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Paraffin embedded block of colorectal carcinoma obtained after biopsy or surgery
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients with colorectal carcinoma: Patient with colorectal carcinoma operated in Martinique between January 1st, 2007 and December 31st, 2009

SUMMARY:
* There is no data at present concerning the KRAS mutation in patients from Martinique with colorectal cancer. Despite the fact that the incidence of this disease continues to increase there is no recent data to confirm it. This study has a descriptive purpose, allowing a comparison of the population from Martinique to other populations.
* A study of incidence of colorectal cancer, overseen by the Association from Martinique for the Epidemiological Search on Cancer (AMREC), also leads to a better knowledge of the local characteristics of the colorectal cancer.
* These two descriptive characteristics of colorectal cancer in Martinique will be useful data for the health professionals to provide their patients better care.

DETAILED DESCRIPTION:
* The colorectal carcinogenesis is complex. It influences among others, the EGFR (Epidermal Growth Factor Receptor) which activation leads to tumoral proliferation, differentiation and invasion. The binding of the EGF (Epidermal Growth Factor) or of another ligand to the EGFR is responsible for the activation of the Ras- Raf and Pi3k pathways.
* The mutation of the genes KRAS, BRAF or PIK3CA results in their continuous activation, independently of the activation or of the pharmacological blocking of EGFR. The most frequently found mutation affects the KRAS gene (20 to 50 % of the cases). 90 % of these mutations are situated on codons 12 and 13 of this gene (70 % codon 12 and 30 % codon 13). These mutations are responsible for a decrease of the GTPase activity of the ras protein, which stays then in active conformation bound to the GTP. This leads to the blocking of the pathway and to the inactivity of the pharmacological blocking of EGFR.

ELIGIBILITY:
Inclusion Criteria:

* for the study of the KRAS mutation: 250 patients drawn by lots among the cases of colorectal carcinoma diagnosed between January 1st, 2007 and December 31st, 2009 in Martinique
* for the study of incidence: patient for whom was diagnosed a colorectal carcinoma between January 1st, 2007 and December 31st, 2009
* patient unopposed and in free agreement to participate in this study
* patient having his main home in Martinique at the time of the diagnosis
* patient 18 years old and over

Exclusion Criteria:

* patient whose diagnosis is prior to 2007 and later in 2009
* patient having shown opposition to the participation in this study
* patient minor or under guardianship
* patient not having his main home in Martinique at the time of the diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who lived in martinique (a french west-indies island) with a colorectal carcinoma diagnosed between january 1st, 2007 and december 31st, 2009
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2011-07; Primary Completion 2011-10 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Frequency of KRAS mutation | 4 months
  Estimate the frequency of the KRAS mutation detected in paraffin embedded blocks of colorectal carcinoma operated in Martinique between 2007 and 2009

SECONDARY OUTCOMES:
The incidence of the colorectal carcinoma | 4 months
  Estimate the incidence of the colorectal carcinoma in Martinique between 2007 and 2009.

CONTACTS AND LOCATIONS:
Overall Officials: Odile BERA, MD, Principal Investigator — Laboratoire de virologie - Centre Hospitalier Universitaire de Fort de France
Locations (1):
- Laboratoire de Virologie - CHU de Fort de France, Fort de France, Martinique, France